CLINICAL TRIAL: NCT06419452
Title: Effects of Unilateral, Bilateral and Combined Resistance Training on the Speed and Accuracy of the Serve in Youth Tennis Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Ma Xudong, Principal Investigator, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MXudong
Record Dates: First submitted 2024-05-09; First posted 2024-05-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Exercise Training
Keywords: Resistance training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral resistance training (Other): Unilateral resistance training uses ipsilateral limb restricted contractions, in which each limb works independently, moving or opposing a given loading task
  Interventions: Other: Unilateral resistance training programme
- Bilateral resistance training (Other): Bilateral resistance training is the contraction of the same muscle in both limbs, that is, both limbs work together in a coordinated manner to cope with a given loading task
  Interventions: Other: Bilateral resistance training programme
- combined resistance training (Other): Combined unilateral and bilateral forms of resistance training
  Interventions: Other: Combined（UL+BL） resistance training programme

INTERVENTIONS:
Other: Unilateral resistance training programme — A method of training that increases muscle strength and endurance by using external resistance to a unilateral limb or movement.
  Arms: Unilateral resistance training
Other: Bilateral resistance training programme — A training method that increases muscle strength and endurance by using external resistance on both limbs or movements,
  Arms: Bilateral resistance training
Other: Combined（UL+BL） resistance training programme — A method of training that uses limbs or movements to increase muscle strength and endurance by external resistance using unilateral and bilateral combined forms,
  Arms: combined resistance training

SUMMARY:
This study is to explore the effects of unilateral, bilateral and combined resistance training on the serve speed and accuracy of amateur youth tennis players in China. The subjects were young male tennis players aged 16-20 years from four universities in Gansu Province.

The experiment was divided into control group (CG), experiment group 1 (EG1-unilateral group), experiment group 2 (EG2-bilateral group) and experiment group 3 (EG3-combined group). Used to compare the effects of different forms of resistance training on serve speed and accuracy. Previous studies have shown that unilateral and bilateral resistance training can effectively improve strength, power, and speed in athletes (Speirs, et al., 2016; Davo, Jimenez, & Solana,. , 2018), there is still controversy when comparing the advantages and disadvantages of two forms of resistance training (Ramirez-Campillo et al., 2015; Donab and Wall. The results of this study will be expected to be updated in 2022. Unilateral resistance training, bilateral resistance training, and combined unilateral and bilateral resistance training were used as intervention models in this study.

Based on the literature review, the training frequency of this experiment was arranged as 2 times/week, and the total training time was 6 weeks, with a fixed duration of each training session. Each training session lasted a maximum of 60 minutes. In this experiment, the interval between the two weekly training sessions was at least 24 h to prevent subjects from being in a fatigued state in the relevant muscle groups of the body and affecting the experimental level.

DETAILED DESCRIPTION:
backgrounds

Originally known as lawn tennis, tennis originated in France and became official in England. There is evidence that people participating in tennis can provide numerous health benefits. Secondly, tennis is a sport with anaerobic metabolism, supplemented by high-intensity aerobic metabolism, which means that tennis has a great demand for speed, strength and other physical qualities. However, in recent years, China's athletes have been in debt for a long time, resulting in weak basic qualities and lack of special ability, which restricts the development of China's athletes. In order to achieve good sports performance, the training method is very important. In the case of adolescents, where strength is gradually declining, evidence suggests that the implementation of scientific resistance training under perfect supervision can help the development of physical fitness and athletic performance. Secondly, resistance training is mostly focused bilaterally, and the advantage of unilateral resistance training is that it is superior to the BLD effect to improve strength than bilateral training. Evidence suggests that isometric strength gains after unilateral resistance training are almost twice as high as those after bilateral resistance training.

Problem statement

Strength levels in today's youth are declining, and evidence suggests that traditional training in youth focuses on bilateral and ignores movement patterns and focuses on single joints, resulting in low stroke power and poor speed in youth tennis players. Existing tennis training has focused on bilateral resistance training or tennis-specific technique training, but the results have not been significant. Tennis serve is very important, and it is the key to win in tennis matches. Evidence shows that muscle strength and explosive power are significantly related to tennis serve. Therefore, it is important to focus on the effects of different resistance training on tennis serve. Secondly, unilateral training is in line with the sport-specific characteristics and compound resistance training is significant for strength as well as explosive power, so these two training modalities are crucial for tennis. To summarize the problem statement of this study, there are three main problem statements, firstly, the importance of serve technique in tennis program, secondly, unilateral training is in line with the specific characteristics of unilateral movement of tennis serve, and thirdly, the importance of combined resistance training in tennis.

Proposed solution Different forms of resistance training will provide different benefits to the athlete, and the sport of tennis is consistent with unilateral movement, in order to achieve better athletic performance as well as skill performance. The researcher will perform the following manipulation.

Provide different forms of resistance training (unilateral, bilateral, and combined) and observe the changes in the athletic performance of tennis players in terms of strength, explosiveness, flexibility, and coordination.

Provide different forms of resistance training (unilateral, bilateral, and combined) and observe the changes in the tennis players' serve speed and serve accuracy

Literature review

This chapter provides detailed information on the relevant literature and contributes to a comprehensive understanding of the following areas: (1) tennis serve characteristics, (2) youth resistance training safety, (3) resistance training programmes and guidelines, (4) youth resistance training and sports performance, (5 ) physical demands of the tennis serve, (6) the importance of unilateral resistance training, (7) the BLD effect of bilateral resistance training, and (8) the validity of combined resistance training. The literature review is concluded with a summary of the literature review.

The work of this study and the outlook

In the available studies, gains from unilateral resistance training and bilateral resistance training appear to produce relatively contradictory results.According to the principle of specificity of training, the structure pattern of training should imitate motor technique structure as much as possible. For example, tennis serving, soccer shooting, badminton spiking and other sports that are presented in the form of unilateral should be intervened by unilateral resistance training.However, bilateral resistance training programmes are widely used in existing studies.Therefore, the aim of this study was to investigate the effect of unilateral and bilateral resistance training on tennis serve performance of a unilateral nature.In addition, the benefits of unilateral and bilateral resistance training in exercise performance such as strength, speed, and explosive power are also different. Studies have shown that unilateral resistance training is more beneficial for exercise performance in the unilateral exercise mode, and bilateral resistance training is more beneficial for exercise performance in the bilateral exercise mode.Some studies, however, have yielded conflicting results. Gonzalo studied 22 male basketball players who completed unilateral and bilateral resistance training on Saturday and found that the unilateral group performed better in the bilateral CMJ than the bilateral group (UL: 37.4 ± 4.2 VS 39.8 ± 5.1, ES=0.47, %∆=6.5; BL: 38.9 ± 5.3 VS 40.6 ± 5.5 ES=0.27, %∆=4.5)In addition, another study showed that unilateral and bilateral resistance training were equally effective in improving lower limb strength in athletes, but there was no significant difference between the two groups (BL:75 ± 4.5 VS 81 ± 4.3; UL:76 ± 6.1 VS 83 ± 5.1, p<0.05).In summary, this study will further confirm the improvement of unilateral and bilateral resistance training in strength, explosive power, coordination and other sports performance.In addition, as unilateral resistance training or reduced stability in unilateral testing has the potential to sacrifice strength development, this study will also focus on the effects of unilateral and bilateral resistance training on bilaterally dominant motor performance such as strength and explosiveness, as well as unilateral pattern tennis serve performance.This will address the occurrence of bilateral sets that are unfamiliar with unilateral training leading to the phenomenon of sacrificing strength to maintain stability.

The phenomenon of migration of athletic performance such as strength and explosiveness in both uni- and multi-joint muscles has been confirmed by numerous studies,but there is little research on the phenomenon of complex skill transfer.This study will determine the effects of unilateral and bilateral resistance training on serving performance, thereby determining if there is also cross-education in complex motor skill performance.In addition, many studies have focused on the effects of unilateral and bilateral resistance training on the lower limbs, so this study will use the upper limb test as one of the indicators.Tennis serve is a complex movement involving multiple joint muscles, which is a process of transforming potential energy stored in the lower limbs into kinetic energy generated in the upper limbs, so the testing of upper and lower limb strength and explosive force indexes is particularly important.

ELIGIBILITY:
Inclusion Criteria:

1. Between 16 and 20 years of age.
2. National second-level athletes or above, or have participated in provincial or municipal competitions, or students majoring in tennis.
3. At least 2 years of tennis training experience.

Exclusion Criteria:

1. Have performed systematic resistance training within the past three months.
2. Medical problems that may affect the study results, including athletes with recent history of surgery or injury.
3. Athletes at high risk for sports injuries.

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Strength | 6 weeks
  Muscle strength is the force produced by a muscle or muscle fibre against resistance
Power | 6 weeks
  Power is the capacity to produce maximum force in a brief time frame
Flexibility | 6 weeks
  Flexibility refers to muscle flexibility and joint mobility, such as the ability of a joint or muscle to move within an unrestricted, non-painful range of motion and to contract
Coordination | 6 weeks
  Coordination is the ability of the body to control muscle groups at the right time, in the right direction and at the right speed, and to mobilise muscles effectively to achieve precise movements
Serve speed | 6 weeks
  Speed is a form of physical quality, which refers to the ability of the human body to move under the specified conditions
Serve accuracy | 6 weeks
  The degree of agreement between the test result and the accepted reference value, understood in the context of tennis as the amount of times the ball moves into the effective target range

CONTACTS AND LOCATIONS:
Locations (1):
- Northwest Normal University, Lanzhou, Gansu, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT06419452/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT06419452/ICF_001.pdf